CLINICAL TRIAL: NCT02314715
Title: Neuromuscular Control in Knee Osteoarthritis
Acronym: NEKO
Status: Completed | Type: Observational
Sponsor: Martijn Steultjens (Other)
Responsible Party: Sponsor-Investigator, Martijn Steultjens, Professor of Musculoskeletal Health, Glasgow Caledonian University
Organization: Glasgow Caledonian University (Other)
Other Study IDs: GCU_MSK_SS_001
Record Dates: First submitted 2014-12-02; First posted 2014-12-11 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2015-03

CONDITIONS: Osteoarthritis Knee
Keywords: Osteoarthritis Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- Knee Osteoarthritis: Participants with diagnosed knee osteoarthritis
- Controls: Participants without knee osteoarthritis

SUMMARY:
Arthritis is one of the most prevailing causes of disability with knee osteoarthritis (KOA) the most common form. The lifetime risk of developing symptomatic KOA by the age of 85 years is 44.7%, where females are at a greater risk (1.8 times) than male counter parts. KOA is the leading cause of limitations in activities of daily living such as walking and climbing stairs particularly in the elderly. This is primarily due to pain and instability of the joint resulting in buckling of knees caused by muscle weakness, joint stiffness and damage. Patients with KOA have larger variations in muscle strength and are unable to maintain a target force combined with impaired ability to perceive joint movement and positioning suggests impaired neuromuscular control (NC) may influence KOA. NC refers to the nervous system's control over muscle activation contributing to task performance. This study aims to establish the role of loss of NC in biomechanical determinants and health outcomes of KOA.

ELIGIBILITY:
Inclusion Criteria:

Knee osteoarthritis participants only:

* Knee Osteoarthritis confirmed by a physician using the American College of Rheumatology (ACR 1986) Criteria
* Have unilateral or bilateral knee osteoarthritis
* Aged 40 years or over.

Healthy control participants only:

* Have no history of unilateral/bilateral knee osteoarthritis
* Had no current chronic/stable knee pain in the past 3 months
* Aged 40 years or over.

Exclusion Criteria:

All participants are excluded if they:

* Have neuromuscular skeletal injury/illness (e.g.Multiple Sclerosis, Parkinson's disease, Muscular Dystrophy, Cerebral Palsy)
* Have had knee surgery, knee arthroplastic surgery and arthroscopic debridement or corrective surgery for knee osteoarthritis in the past 12 months
* Have had corticosteroid injections to or around the knee in the past 3 months.
* Have unstable heart disease
* Previously had a stroke
* Have insulin-dependent diabetes
* Have osteoporosis
* Have a history of falls and other motor deficits
* Are unable to walk up and down stairs
* Are unable to rise from a chair without the aid of another person
* Have an unstable medication schedule and medication that causes dizziness
* Have Dementia/Alzheimer's/ an inability to comprehend, follow instructions and give informed consent
* Have an inability to lie flat for 60 minutes Have mental in their body.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary and secondary care clinics, and general community.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2013-11; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Neuromuscular Control | 1 day
  Neuromuscular control will be assessed through muscle co-activation index from electromyography (EMG) of the hamstrings, quadriceps and gastrocnemius. The electromechanical delay (delay between the onset of EMG and force), active proprioception and force accuracy and steadiness measure determined from submaximal isometric contractions will be used to determine neuromuscular control

SECONDARY OUTCOMES:
Disease Outcome | 1 day
  Joint damage scored using the Boston Leeds Osteoarthritis Knee Score (BLOKS) from 1.5T MRI along with pain and function assessed from knee injury and osteoarthritis score (KOOS) and patient reported outcomes measurement information system (PROMIS) will be used to determine disease outcome.

OTHER OUTCOMES:
Determinants of knee osteoarthritis | 1 day
  Muscle strength (peak force) will be assessed from maximal isometric contractions of the knee, along with passive motion and position sense proprioception as determinants of knee osteoarthritis.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie L Smith, MRes, Principal Investigator — Glasgow Caledonian University
Locations (1):
- Glasgow Caledonian University, Glasgow, United Kingdom

REFERENCES:
- [Derived] Smith SL, Allan R, Marreiros SP, Woodburn J, Steultjens MPM. Muscle Co-Activation Across Activities of Daily Living in Individuals With Knee Osteoarthritis. Arthritis Care Res (Hoboken). 2019 May;71(5):651-660. doi: 10.1002/acr.23688. PMID 29953745